CLINICAL TRIAL: NCT01641653
Title: Does the Administration of Preop Midazolam Assist in Maintaining Blood Glucose Norms in Non-diabetic Patient During the Perioperative Period
Brief Title: Does Preop Midazolam Maintain Blood Glucose Norms in the Non Diabetic Perioperative Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120110037
Record Dates: First submitted 2011-12-08; First posted 2012-07-17 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2014-11

CONDITIONS: Hernia
Keywords: Nondiabetics undergoing hernia repair.
MeSH Terms: conditions — Hernia | interventions — Saline Solution; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): half of the patients will receive placebo (normal saline 2cc/) prior to entering the OR
  Interventions: Other: Normal saline
- Midazolam (Active Comparator): half of the patients will receive Midazolam 1-2.5mg prior to entering the OR
  Interventions: Drug: Midazolam

INTERVENTIONS:
Other: Normal saline — Normal saline 2cc. one dose prior to OR
  Arms: placebo
Drug: Midazolam — 1-2.5 mg
  Other Names: Versed
  Arms: Midazolam

SUMMARY:
This research is being done to investigate if patients who receive a commonly used sedative drug, known as midazolam, are likely to have high blood sugar levels during the stressful period during and immediately after surgery. A sedative drug is used to relax a person without making them sleepy. This drug is also helpful in reducing the memory of the stressful experience before the anesthesiologists administers anesthesia. Everyone has glucose or sugar in their blood stream. This sugar gives energy to our organs to allow them to work. Since high blood sugar levels may be associated with complications like wound infections, the investigators research is being done to find if patients who receive a sedative medication prior to their surgical procedure have lower blood sugars during the surgery then a patient who does not receive the sedation. The investigators would like to know if the administration of this commonly used drug will help patients maintain a normal glucose level during a stressful period.

DETAILED DESCRIPTION:
Surgery performed during general anesthesia induces a stress response partially through a catabolic energy state. As a result, serum glucose may rise to levels which have been associated with major morbidity and mortality. In patients undergoing cardiac surgery, typically "tight glycemic control" strategies are used to prevent hyper- and hypo-glycemia in the perioperative period, before the effects of perioperative hyperglycemia begin to emerge. In one study a high percentage of patients in the control group had intraoperative blood glucose levels over 225. After one hour of surgery: 20%, after two hours: 28%, after three hours: 31% and in the post-anesthesia recovery room: 52% of patients. These high levels of glucose could be associated with significant post-operative morbidity such as wound infection and pneumonia as shown in the cardiac surgery population.

Glucose alterations induced by psychological stress have been studied in rats but not in humans.

Midazolam is a short acting benzodiazepine that depresses central nervous system. It is indicated for anxiolysis, amnesia and sedation. We hypothesize that the administration of midazolam may be beneficial in suppressing the catabolic energy state, maintaining normal glucose levels during this stressful period. This commonly available inexpensive drug, which is tolerated well by the majority of patients, may be useful in maintaining normal glucose levels and minimize adverse postoperative outcomes, such as wound and urinary tract infections and pneumonia.

We propose a prospective, single blind (subject only) randomized study to measure glucose levels in non diabetic patients undergoing both ventral and inguinal hernia repair. Patients scheduled for hernia repair will be approached on the morning of surgery (on E yellow) and following the completion of the informed consent process, a preoperative capillary glucose reading will be performed via the portable Abbott Freestyle™ Glucometer. Subjects with a preoperative reading of greater than 110 will be excluded from the study. Prior to the administration of any medication, we will ask all subjects to complete the State Trait Anxiety Inventory for Adults (STAI Form Y-1 and Y-2). This is a research instrument for anxiety in adults. It is comprised of 40 questions at a 6th grade reading level. It is designed to differentiate between the temporary condition of "state anxiety" and a long term personality trait. We will determine whether the subjects' perioperative glucose level correlates with the his/her score on the STAI.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic preoperative fasting blood sugar level of 110 mg/dL or less.

Exclusion Criteria:

* Fasting blood sugar > than 110mg/dL
* Subjects who are pregnant
* Subjects who do not speak English
* Subjects who are on steroids prior to admission
* Hypersensitivity to midazolam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Tilak, MD, Principal Investigator — UMDNJ/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6/21/11-8/9/12 preoperative holding area
Pre-assignment Details: Non diabetics with fasting blood sugar < = to 110mg/dL scheduled for an elective hernia repair
Groups:
- Placebo: half of the patients will receive placebo (normal saline 2mL) prior to entering the OR
  Normal saline: Normal saline 2cc. one dose prior to OR
- Midazolam: half of the patients will receive Midazolam prior to entering the OR
  Midazolam: 1-2.5 mg
Period: Overall Study
Arm/Group | Placebo | Midazolam
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: non diabetics undergoing hernia repair
Groups:
- Placebo: half of the patients will receive placebo (normal saline) prior to entering the OR
  Normal saline: Normal saline 2cc. one dose prior to OR
- Total: Total of all reporting groups
Arm/Group | Placebo | Midazolam | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 21 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants] — participants scheduled for hernia repair were screened and consented, preoperative glucose level was then performed with Abbott Freestyle monitor to insure that fasting glucose level was below or equal to 110mg/dL.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 13 | 11 | 24
    White | 9 | 12 | 21
    More than one race | 2 | 3 | 5
    Unknown or Not Reported | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Maximum Perioperative Blood Glucose Level of 30 Minute Interval Measurements
Description: Non diabetic subjects undergoing hernia repair were randomized into 2 groups. Midazolam vs. placebo. Blood glucose level was monitored preoperatively and following induction of anesthesia at 30 minute intervals perioperatively, and after in the PACU at 30 minutes and 60 minutes following arrival. All readings were performed using the Abbott Freestyle Glucose Monitor.
Time Frame: every 30 min for duration of surgery
Population: per protocol
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Placebo: Normal saline: Normal saline 2cc. IV one dose prior to OR
- Midazolam: One half of subjects will recieveMidazolam: 1-2.5 mg IV
Arm/Group | Placebo | Midazolam
Number analyzed (Participants) | 30 | 30
mg/dL | 114.0 [101.0 to 126.0] | 108.0 [101.0 to 125.0]
Statistical Analysis 1: Comparison: Placebo vs Midazolam; This is a pilot study no power calculation was performed. The Wilcoxon rank-sum test was used to assess differences in max intraop glucose between placebo and midazolam groups; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Glucose Level Percent Change From Pre-op to Maximum Glucose Level
Description: blood glucose level measured preoperatively, through surgical period and in PACU at 30 min and 60 min
Time Frame: Preoperatively, intraoperatively 30 min for duration of surgery
Population: per protocol
Measure: Median (Inter-Quartile Range); unit: percentage of increase in glucose level
Groups:
- Midazolam: half of subjects will receive Midazolam: 1-2.5 mgIV prior to entering the OR
Arm/Group | Placebo | Midazolam
Number analyzed (Participants) | 30 | 30
percentage of increase in glucose level | 24.9 [10.99 to 38.10] | 14.9 [7.69 to 37.50]
Statistical Analysis 1: Comparison: Placebo vs Midazolam; percent change in glucose levels from preoperative level to maximum perioperative measurement level; Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 10

3. Secondary Outcome: Percent Intra-op Blood Glucose Level of 140mg/dL or Less
Description: blood glucose level will be tested perioperatively at 30 minute intervals following induction. All glucose levels will be recorded .midazolam group will maintain a blood glucose level perioperatively of 140mg/dL or less
Time Frame: perioperatively
Measure: Number; unit: percentage of glucose levels<140
Groups:
- Placebo: subjects will receive 2cc. Normal Saline prior to entering the OR
- Midazolam: subjects will receive midazolam 1.5-2mg prior to entering the OR
Arm/Group | Placebo | Midazolam
Number analyzed (Participants) | 30 | 26
percentage of glucose levels<140 | 100 | 86.6
Statistical Analysis 1: Comparison: Placebo vs Midazolam; Test type: Superiority or Other; p = 0.12, Chi-squared, Corrected — Chi-square with continuity correction

ADVERSE EVENTS:
Arm/Group | Placebo | Midazolam
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes